CLINICAL TRIAL: NCT02631200
Title: Advance Care Planning With Older Patients Who Have End-stage Kidney Disease: Feasibility of a Deferred Entry Randomised Controlled Trial Incorporating a Mixed Methods Process Evaluation
Brief Title: Advance Care Planning With Older Patients Who Have End-stage Kidney Disease
Acronym: ACREDiT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Queen's University, Belfast (Other)
Collaborators: The Dunhill Medical Trust (Other)
Responsible Party: Principal Investigator, Peter O'Halloran, Dr, Queen's University, Belfast
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 20724-1
Record Dates: First submitted 2015-10-28; First posted 2015-12-16 (Estimated); Results first posted 2024-07-29 (Actual); Last update posted 2024-07-29 (Actual); Status verified 2024-02

CONDITIONS: Kidney Failure, Chronic
Keywords: Advance Care Planning; Palliative care; Frail Elderly; Renal Dialysis
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Advance care plan (Experimental): Participants will be offered the opportunity to complete an advance care plan.
  Interventions: Behavioral: Advance care plan
- Usual care (No Intervention): Participants will be offered usual care for 12 weeks (and only then be offered the opportunity to complete an advance care plan).

INTERVENTIONS:
Behavioral: Advance care plan — Participants will be offered the opportunity to complete an ACP by a nurse trained as an ACP facilitator, who will discuss the process with them using standard materials. At least 48 hours later, they will complete an ACP document with the help of the ACP facilitator, working together with trained expert patients who will provide peer support at the time of ACP completion and subsequently by telephone, assisted where necessary by the ACP facilitator.
  Arms: Advance care plan

SUMMARY:
This study will test the feasibility of carrying out a randomised controlled trial, incorporating a mixed methods process evaluation, to evaluate advance care planning with older patients who have end-stage kidney disease.

DETAILED DESCRIPTION:
Kidney failure becomes more common as people age. It increases the risks of other major illnesses, sudden worsening of symptoms, and death. Even so, many people with kidney failure do not talk about their preferences for end-of-life care.

Advance care planning (ACP) can help patients and families think through their preferences for future care and discuss these with the professionals looking after them. This may lead to care more in keeping with patients' wishes and so reduce distress for patients and families. ACP is recommended as good practice for people with kidney failure.

However, questions remain about the impact of ACP on patients and families; and also about the best ways to put ACP into practice. Doing research about ACP is challenging for everyone involved, so we need to thoroughly test our research methods in a pilot study before we attempt a larger study that would fully answer those questions.

To test our methods we will carry out a small-scale randomised controlled trial comparing those patients who use ACP with those who do not, in terms of: quality of life, anxiety, depression, physical functioning, well-being, satisfaction with decision-making and agreement between the patient and their nominated carer in terms of the patient's preferences for care at the end of life.

ELIGIBILITY:
Inclusion Criteria:

* Attending the renal units taking part in the study
* Receiving renal replacement therapy
* Capacity to understand, retain, and weigh the necessary information and communicate their decisions
* Identified by their consultant as having worsening symptoms, functional decline, and two or more co-morbidities.

Exclusion Criteria:

* Expected to die in the next three months

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 36 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2018-07 (Actual); Study Completion 2018-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter D O'Halloran, PhD, Principal Investigator — Queen's University, Belfast
Locations (1):
- Queen's University Belfast, Belfast, Northern Ireland, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Deidentified data that underlie the results reported in this article are available to qualified researchers for approved scientific uses immediately following publication of the trial results* with no end date. Data access proposals should be directed to the corresponding author. The Trial Protocol is available on request.
  *DOI https://doi.org/10.1186/s12882-020-02129-5
Supporting Information: Study Protocol
Time Frame: Immediately following publication of the trial results* with no end date.
  *DOI https://doi.org/10.1186/s12882-020-02129-5
Access Criteria: Available to qualified researchers for approved scientific uses.
URL: https://doi.org/10.1186/s12882-020-02129-5

REFERENCES:
- [Derived] O'Halloran P, Noble H, Norwood K, Maxwell P, Murtagh F, Shields J, Mullan R, Matthews M, Cardwell C, Clarke M, Morton R, Shah K, Forbes T, Brazil K. Nurse-led advance care planning with older people who have end-stage kidney disease: feasibility of a deferred entry randomised controlled trial incorporating an economic evaluation and mixed methods process evaluation (ACReDiT). BMC Nephrol. 2020 Nov 13;21(1):478. doi: 10.1186/s12882-020-02129-5. PMID 33187506

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment began in December 2016 and lasted 189 days. Participants were recruited from two haemodialysis units in Northern Ireland, UK. Nephrologists approached patients and those interested were given patient information packs for themselves and a surrogate. The ACP nurse returned to the patient 2-7 days later to seek their consent. Surrogates could contact the research team directly using a dedicated phone number or email address, or a form and reply-paid envelope
Period: First Period
Arm/Group | Advance Care Plan | Usual Care
Started | 17 | 19
Completed | 10 | 12
Not Completed | 7 | 7
Not completed — Death | 1 | 2
Not completed — Patient ill-health | 2 | 4
Not completed — Withdrawal by Subject | 4 | 1
Period: Deferred Period
Arm/Group | Advance Care Plan | Usual Care
Started (This was a deferred entry randomised controlled trial in which patients and their nominated surrogate were allocated in a 1:1 ratio to either immediate or deferred entry groups. Participants in the deferred entry group had outcomes measured contemporaneously with the immediate entry group but received the intervention 12 weeks after baseline data collection. They were then followed up until 24 weeks.) | 0 | 12
Completed | 0 | 7
Not Completed | 0 | 5
Not completed — Death | 0 | 1
Not completed — Received kidney transplant | 0 | 1
Not completed — Withdrawal by Subject | 0 | 2
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Advance Care Plan | Usual Care | Total
Number analyzed (Participants) | 17 | 19 | 36
Age, Continuous [Mean (Standard Deviation); unit: years] | 75.6 (6.81) | 73.2 (5.01) | 74.9 (6.89)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 6
  Male | 14 | 16 | 30
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 17 | 19 | 36
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United Kingdom | 17 | 19 | 36

OUTCOME MEASURES:

1. Primary Outcome: Kidney Disease Quality
Description: Quality of life as measured by the Kidney Disease Quality of Life instrument - Short Form (KDQOL-36™). The KDQOL-36 has five scales, including two generic health related quality of life (HRQOL) scales from the Short-Form (SF)-12 version 1 (12 items total) and three kidney-specific scales (24 items total). Each scale has a minimum score of zero and a maximum of 100. Higher scores reflect better quality of life and a better outcome. Subscales are not combined.
Time Frame: 12 weeks post intervention
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Advance Care Plan | Usual Care
Number analyzed (Participants) | 10 | 12
score on a scale
  KDQOL-36™ - Symptoms | 75.4 (13.3) | 78.3 (19.2)
  KDQOL-36™ - Effects | 78.4 (16.0) | 73.4 (21.6)
  KDQOL-36™ - Burden | 46.9 (23.8) | 55.2 (25.7)
  SF12 physical | 31.5 (9.5) | 34.9 (13.0)
  SF12 mental | 53.3 (6.9) | 52.4 (6.9)

2. Secondary Outcome: Number of Participants With Agreement Between the Patient and Their Nominated Carer in Terms of the Patient's Preferences
Description: Number of Participants with Agreement between the patient and their nominated carer in terms of the patient's preferences. We will measure this by asking the carer to make an independent assessment of the patient's preferences in relation to the key information covered by the ACP intervention, before taking part in the ACP.
Time Frame: 12 weeks post intervention
Measure: Count of Participants; unit: Participants
Arm/Group | Advance Care Plan | Usual Care
Number analyzed (Participants) | 17 | 19
Participants
  Surrogate named | 10 | 7
  Surrogate not named | 7 | 12
  Surrogate participated | 7 | 3
  Surrogate did not participate | 3 | 4
  Surrogate's understanding of ACP converged with patient's on at least one dimension of ACP | 3 | 0
  Surrogate's understanding of ACP did not converged with patient's | 4 | 3

3. Secondary Outcome: Depression
Description: Degree of anxiety, depression, well-being, functioning and risk as measured by the Clinical Outcomes in Routine Evaluation measure (CORE 34) a 34- item Likert-type scale scored on a 5-point scale ranging from 0 (not at all) to 4 (most or all the time). The minimum mean value is zero and the maximum is 4. Higher scores indicate greater distress and a worse outcome. Mean scores from reference groups are 1.86 (SD 0.75) for those referred to psychiatric services and 0.76 (SD 0.59) for the general population.
Time Frame: 12 weeks post intervention
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Advance Care Plan | Usual Care
Number analyzed (Participants) | 10 | 12
score on a scale | 0.4 (0.3) | 0.4 (0.3)

4. Secondary Outcome: The Degree to Which the Patient Felt That They Had Shared in Decision-making.
Description: The degree to which the patient felt that they had shared in decision-making about their care as measured by the Patient Experience of Shared Decision Making (SHARED) instrument. This is a a ten-item Likert-type scale ranging from 'Disagree strongly' to 'Agree strongly', with one point for 'Agree', two for 'Agree strongly', and no points for disagreement. The minimum score is zero and the maximum is 20. Higher scores indicate more sharing and a better outcome.
Time Frame: 12 weeks post intervention
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Advance Care Plan | Usual Care
Number analyzed (Participants) | 2 | 6
score on a scale | 12 (5.7) | 11.2 (6.0)

ADVERSE EVENTS:
Time Frame: 15 months.
Arm/Group | Advance Care Plan | Usual Care
All-Cause Mortality (participants affected / at risk) | 1/17 | 3/19
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/19
Other Adverse Events (participants affected / at risk) | 0/17 | 0/19

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2017-01-30): https://cdn.clinicaltrials.gov/large-docs/00/NCT02631200/Prot_SAP_000.pdf
  • Informed Consent Form (2016-01-04): https://cdn.clinicaltrials.gov/large-docs/00/NCT02631200/ICF_001.pdf